CLINICAL TRIAL: NCT01844154
Title: Fracture and Fall Prevention in Elderly With Osteoporosis: Long-term Follow up
Brief Title: Fracture and Fall Prevention in Elderly With Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201204059RIC
Record Dates: First submitted 2012-10-05; First posted 2013-05-01 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Osteoporosis, Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Osteoporosis is a prevalent health concern among older adults and is associated with an increased risk of falls that can cause fracture, injury or mortality. Identifying the factors related to falls occurring within this population is essential for the development of effective regimes for fall prevention. Studies have shown that muscle quality and good posture alignments are critical for balance control in older adults. People are diagnosed with osteoporosis often combining with muscles weakness, and increased spine kyphosis leading vertebral, fractures and poor balance control, even falls. Therefore, improving muscle quality, strengthening weak muscles and correcting postural alignment are essential elements for fracture and fall prevention in older adults with osteoporosis. The long-term objectives of this work are to prevent fracture and fall in older adults with osteoporosis by improving the function of degenerative muscles using exercise training.

ELIGIBILITY:
osteopenia or osteoporosis group:

Inclusion Criteria:

* able to stand and walk for 5 minutes independently
* having normal or corrected to normal vision
* having age between > 50 years
* already have DEXA and X-ray exam with osteopenia (-2.5 < t-score < -1.0) or osteoporosis (t-score <-2.5)

Exclusion Criteria:

* being pregnant
* sensory-motor deficits
* inability of communication
* lack of access to a telephone
* t-score <-2.5 combine with existing fracture

control age-matched group:

Inclusion Criteria:

* able to stand and walk for 5 minutes independently
* having normal or corrected to normal vision
* having age between > 50 years
* already have DEXA and X-ray exam without osteopenia or osteoporosis (t-score > -1.0)

Exclusion Criteria:

* being pregnant
* sensory-motor deficits
* inability of communication
* lack of access to a telephone
* t-score <-2.5 combine with existing fracture

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: osteopenia (-2.5 < t-score < -1.0) or osteoporosis (t-score <-2.5)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Muscle activation during balance recovery | every 3 month, up to 1 year
  Data collection will be carried out in 2 sessions in 2 different days within the span of a week. The first day of data collection includes basic information, anthropometric measure, clinical tests, and functional tests. The second day of data collection includes muscle and joint assessment, and biomechanical tests. Each session last approximately 2.5 hours in duration.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PT,PhD, Principal Investigator — School of physical therapy, National Taiwan University
Locations (2):
- Taiwan (2):
  - National Taiwan University, Taipei, Taiwan
  - School & Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei